CLINICAL TRIAL: NCT05466006
Title: Peri-implant Soft Tissue Volume Changes After Treatment of Small Buccal Dehiscence With Volume-stable Collagen Matrix or Connective Tissue Graft: a Randomized Controlled Clinical Trial
Brief Title: Peri-implant Soft Tissue Volume Changes at Small Buccal Dehiscences
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mario Aimetti, Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFGTurin2
Record Dates: First submitted 2022-07-08; First posted 2022-07-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Dental Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subepithelial Connective Tissue Graft (SCTG) (Active Comparator): Soft tissue augmentation at peri-implant small buccal dehiscence with subepithelial connective tissue graft harvested from the patient's palate
  Interventions: Procedure: Soft tissue augmentation with subepithelial connective tissue graft (SCTG)
- Volume Stable Collagen Matrix (VCMX) (Experimental): Soft tissue augmentation at peri-implant small buccal dehiscence with xenogenic volume stable collagen matrix
  Interventions: Procedure: Soft tissue augmentation with xenogenic volume stable collagen matrix (VCXM)

INTERVENTIONS:
Procedure: Soft tissue augmentation with subepithelial connective tissue graft (SCTG) — After the assessment of the vestibular bone dehiscence at implant site from the most apical extension of the trans-mucosal implant collar (≤3 mm evaluated in a vertical direction), SCTG will be harvested from the palate and sutured to the flap. Simple interdental sutures will be performed in order to stabilize the flap in close contact with the healing screw.
  Arms: Subepithelial Connective Tissue Graft (SCTG)
Procedure: Soft tissue augmentation with xenogenic volume stable collagen matrix (VCXM) — After the assessment of the vestibular bone dehiscence at implant site from the most apical extension of the trans-mucosal implant collar (≤3 mm evaluated in a vertical direction), VCMX will be sutured to the flap and simple interdental sutures will be performed in order to stabilize the flap in close contact with the healing screw.
  Arms: Volume Stable Collagen Matrix (VCMX)

SUMMARY:
This study was designed to assess peri-implant soft tissue health, volume and marginal stability at implants sites which presented small buccal bone dehiscences (<3mm evaluated in a vertical direction) at the time of insertion. Patients will be then randomly allocated to receive grafting with connective tissue graft or volume stable collagen matrix and evaluated at 3 months after surgery and at 12 months of follow up after crown placement.

ELIGIBILITY:
Inclusion Criteria:

* Single tooth edentulous space
* Expected small buccal bone dehiscence (≤3mm evaluated in a vertical direction) assessed according to the prosthetically guided position of an implant of 4 mm in diameter planned using the pre-surgical CBCT
* Completed non-surgical periodontal therapy (if needed)
* FMPS and FMBS < 20%

Exclusion Criteria:

* Age < 18 years old
* Pregnancy or lactation
* Heavy smokers (> 10 cigarette/day)
* Conditions or diseases contraindicating surgical interventions
* Absence of the expected small buccal bone dehiscence (≤3mm evaluated in a vertical direction) verified after implant placement
* Need for bone regeneration at the implant site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric buccal soft tissue changes (-5 to +5 mm with positive values representing an increase in volume) | 12 months
  Mean linear change in mm at the buccal aspect 1mm below the soft tissue margin
Change in Buccal Probing Pocket Depth (PD) at implant site (0-15 mm with higher values representing worse outcomes) | 12 months
  The distance between the buccal soft tissue margin and the base of the pocket
Mucosal recession at the buccal aspect of the implant site (0-15 mm with higher values indicating worse outcomes) | 12 months
  The distance between the crown margin and the mucosal margin
Pain (VAS scale)(0-10 with higher values indicating worse outcomes) | 12 months
  Subjective pain experienced by the patient expressed in a VAS scale
Bleeding on probing (0 no bleeding, 1 presence of bleeding) | 12 months
  Bleeding after probing within 15 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy

REFERENCES:
- [Derived] Ferrarotti F, Baima G, Mohammadi G, Carboncini C, Romano F, Aimetti M. Peri-Implant Soft Tissue Increase at Small Buccal Bone Dehiscences With Either Volume-Stable Collagen Matrix or Connective Tissue Graft: A Randomized Controlled Trial. Clin Oral Implants Res. 2025 Jul;36(7):846-858. doi: 10.1111/clr.14430. Epub 2025 Mar 19. PMID 40105088